CLINICAL TRIAL: NCT05861063
Title: The Efficacy and Safety of Dezocine Pretreatment for Pain Relief in Acne Scar
Brief Title: The Efficacy and Safety of Dezocine Pretreatment for Pain Relief in Acne Scar Treatment of Fractional CO2 Laser
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: XijingH-PF-20232019-F-1
Record Dates: First submitted 2023-04-17; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-02

CONDITIONS: Acne Atrophica
Keywords: Acne Scar, Dezocine, Pain Relief, Fractional CO2 Laser
MeSH Terms: interventions — dezocine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): The patients were divided into 3 groups based on different dosages of Dezocine injection, with 35 patients in each group: Group 1: Dezocine low-dose group, Group 2: Dezocine high-dose group; Group 3: Blank control group (normal saline).
  Interventions: Device: Fractional CO2 laser
- Dezocine low dose group (Experimental): The patients were divided into 3 groups based on different dosages of Dezocine injection, with 35 patients in each group: Group 1: Dezocine low-dose group, Group 2: Dezocine high-dose group; Group 3: Blank control group (normal saline).
  Interventions: Device: Fractional CO2 laser; Drug: Dezocine
- Dezocine high dose group (Experimental): The patients were divided into 3 groups based on different dosages of Dezocine injection, with 35 patients in each group: Group 1: Dezocine low-dose group, Group 2: Dezocine high-dose group; Group 3: Blank control group (normal saline).
  Interventions: Device: Fractional CO2 laser; Drug: Dezocine

INTERVENTIONS:
Device: Fractional CO2 laser — All patients were given oral administration of 0.5mg paronosetron hydrochloride and lidocaine cream 1 hour before surgery. After cleaning and disinfection, fractional CO2 laser treatment was given. Among them, the fractional CO2 laser laser (American Medical Laser company) selected relatively constant energy parameters in the treatment
  Other Names: paronosetron hydrochloride and lidocaine cream
Drug: Dezocine — Desocine injection was injected intravenously half an hour before surgery (10ml normal saline was added for more than 30 seconds)
  Arms: Dezocine high dose group; Dezocine low dose group

SUMMARY:
The Efficacy and Safety of Dezocine Pretreatment for Pain Relief in Acne Scar Treatment of Fractional CO2 Laser

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old, regardless of gender;
2. Clinical diagnosis of atrophic acne scars;
3. Planning to undergo ultra-pulsed CO2 lattice laser therapy;
4. The patient agrees to participate in this experiment and signs an informed consent form

Exclusion Criteria:

1. Those who take sedative drugs for a long time;
2. Patients with sleep apnea syndrome, previous history of hypertension, and blood pressure greater than 160/100mmHg
3. People with severe heart and lung diseases, liver and kidney diseases, psychosis, pregnancy, and communication disorders;
4. Persons who are known to be allergic to the main drug or any of the excipients in Dezocine injection;
5. Increased intracranial pressure or head injury;
6. Acute and chronic alcoholism;
7. People with hypotension, hypothyroidism, acute episodes of asthma, and epilepsy

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score for Pain | 24 hours
  0 was classified as painless and 10 was classified as unbearable pain. Marks were made on the corresponding parts of the ruler and scores were scored according to the degree of patient's feeling
Hemodynamic parameters | 24 hours
  diastolic blood pressure (DBP), systolic blood pressure (SBP)
Heart rate (HR) | 24 hours
  Hemodynamic parameters
oxygen saturation (SpO2) | 24 hours
  Hemodynamic parameters

SECONDARY OUTCOMES:
Occurrence of Adverse Reactions | 24 hours
  Nausea, vomiting，dizziness，respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No